CLINICAL TRIAL: NCT05218343
Title: Modifying Default Dosing During Electronic Prescribing to Impact Prescribing of High-risk Drugs in Hospitalized Elderly Patients: A Cluster Randomized Controlled Trial With Crossover
Brief Title: An Intuitive, Non-intrusive, Approach to Reduce Patient Harm From Inappropriate Dosing of High-risk Drugs in Older Adult Patients Across an Urban Safety Net Hospital System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Jashvant Poeran, Associate Professor Depts. of Population Health Science & Policy / Orthopedics / Medicine Director, Center for Clinical and Outcomes Research, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: GCO-21-0383
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Potentially Inappropriate Medications
Keywords: Electronic Health Records; Hospital Medication Systems; Geriatrics; Pharmacy; Electronic Prescribing; High-risk drugs

STUDY DESIGN:
Intervention Model Description: This cluster randomized crossover (CRXO) trial involves 10 sites in an urban health system: five clinics will start the trial under the intervention/control during a first time period (T1) then will switch to intervention/control status (T2). The primary outcome is prescription rate of a lower default dose for 8 high-risk drugs.
  Other inputs used for trial design were: baseline rate of prescriptions meeting the geriatric standard (sources: local data, Geriatrics At Your Fingertips), within-period intraclass correlation coefficient (ICC, correlation between two randomly chosen observations in the same cluster), cluster autocorrelation (ratio of between-period ICC to within-period ICC), and coefficient of variation of cluster sizes (required when unequal sample size per cluster is expected). The aim is for ≥80% power to detect a ≥50% increase in prescriptions meeting the geriatric standard; this is based on previous studies and on the researchers' preliminary data on Trazodone.
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers will be unaware of the intervention. However, prescribers will be able to prescribe all available doses, without any restrictions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No change in default dose or frequency selected for the eight targeted drugs
- Intervention (Experimental): The first option a prescriber sees when prescribing any of eight high-risk drugs for elderly hospitalized patients will be modified; the first frequency option a prescriber sees will be modified as well. Providers retain the ability to prescribe any dose or frequency.
  Interventions: Behavioral: EHR-based "nudge" interventions

INTERVENTIONS:
Behavioral: EHR-based "nudge" interventions — Change/introduction of default drug and frequency during electronic prescribing of high-risk drugs for a patient aged ≥65 years
  Arms: Intervention

SUMMARY:
This study will assess whether a modification in the default dose and frequency (the first option a provider sees) during electronic prescribing of a high-risk drug can impact prescribing behavior and subsequent changes in average dose for the targeted high-risk drug, when prescribed to a hospitalized patient aged ≥65 years. In this cluster randomized crossover (CRXO) trial we will randomize a non-intrusive "nudge" intervention, which involves modifying the default dose for high-risk drugs when prescribed electronically to hospitalized patients aged ≥65 years. The CRXO trial involves 10 sites in an urban health system: five sites will start the trial under the intervention/control during a first time period (T1) after which they switch intervention/control status (T2). The primary outcome is prescription rate of a lower default dose (i.e. the geriatric standard) for 8 high-risk drugs. This study will inform the effectiveness of EHR-based "nudge" interventions to reduce inappropriate prescribing of high-risk drugs for elderly patients.

Analyses ongoing, expected to finalize spring 2023

ELIGIBILITY:
Inclusion Criteria:

* a patient must be hospitalized
* 65-years old or older
* receive one of the targeted medications

Exclusion Criteria:

- none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8640 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Prescription rate of modified default dose for eight high-risk drugs | 24 weeks
  Rate at which the modified default dose (geriatric standard) and frequency for eight high-risk drugs are prescribed.

SECONDARY OUTCOMES:
Drug-specific prescription rate | 24 weeks
  Drug-specific prescription rate of the modified default dose for each of the eight high-risk medications and type of order (frequency/type of order).
Mean per-patient dose | 24 weeks
  Mean per-patient dose of the relevant individual high-risk drugs.
Rate of inpatient falls | 24 weeks
  Inpatient falls (with and without injury)
Rate of 30-day readmissions | 30 days post-discharge regarding hospitalization during which a high-risk drug was prescribed
  30-day readmission rates for patients aged ≥65 years who received any of the eight high-risk drugs during their hospitalization.
Length of hospital stay | 24 weeks
  Duration of hospitalization in days for patients aged ≥65 years who received any of the eight high-risk drugs during their hospitalization.
Cost of hospital stay | 24 weeks
  Cost of hospitalization in USD for patients aged ≥65 years who received any of the eight high-risk drugs during their hospitalization.
Spillover effects to patients aged <65 | 24 weeks
  The rate of prescriptions of the newly defaulted (geriatric) dose for any of the eight high-risk drugs among patients aged <65 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jashvant Poeran, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - NYC Health+Hospitals, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Sharing IPD was not something including in the IRB application process. Only aggregated data will be disseminated.